CLINICAL TRIAL: NCT00086242
Title: Stress-Immune Response and Cervical Cancer
Brief Title: Telephone Counseling or Standard Care in Patients Who Have Completed Treatment for Stages I, II, or III Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Lari Wenzel, Professor, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UCIRVINE-2003-3030; CDR0000510143 (Registry Identifier: PDQ (Physician Data Query)); R21CA098794 (NIH)
Record Dates: First submitted 2004-06-28; First posted 2004-06-29 (Estimated); Last update posted 2019-03-08 (Actual); Status verified 2019-03

CONDITIONS: Cervical Cancer; Psychosocial Effects of Cancer and Its Treatment
Keywords: psychosocial effects of cancer and its treatment; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychosocial Telephone Counseling (PTC) (Experimental): Eligible patients are randomized to receive psychosocial telephone counseling (PTC) or usual care.The PTC intervention was specifically designed to help women cope with the stressful events and feelings of distress associated with cervical cancer. The PTC arm of the study received six counseling sessions, ~45 to 50 min in length, in their preferred language, consisting of five consecutive weekly sessions and a 1-month booster session, delivered by a psychologist. A review letter, generated by the counselor after each session, recapitulated the session's contents and reinforced adaptive coping strategies.
  Interventions: Behavioral: Psychosocial Telephone Counseling (PTC)
- Usual Care (No Intervention): Eligible patients are randomized to receive either psychosocial telephone counseling (PTC) or usual care. The usual care are were only contacted by the study team to collect data in an identical frame to subjects receiving PTC.

INTERVENTIONS:
Behavioral: Psychosocial Telephone Counseling (PTC) — Eligible patients are randomized to receive psychosocial telephone counseling (PTC) or usual care.The PTC intervention was specifically designed to help women cope with the stressful events and feelings of distress associated with cervical cancer. The PTC arm of the study received six counseling sessions, ~45 to 50 min in length, in their preferred language, consisting of five consecutive weekly sessions and a 1-month booster session, delivered by a psychologist. A review letter, generated by the counselor after each session, recapitulated the session's contents and reinforced adaptive coping strategies.
  Arms: Psychosocial Telephone Counseling (PTC)

SUMMARY:
RATIONALE: Telephone counseling after treatment may reduce stress and improve the well-being and quality of life of patients who have cervical cancer. Changes in quality of life may be related to changes in immune function and neuroendocrine function.

PURPOSE: This randomized phase I trial is studying how well telephone counseling works compared to standard care in reducing stress in patients who have completed treatment for stage I, stage II, or stage III cervical cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare quality of life (QOL) at baseline and changes in QOL, immune response, and neuroendocrine parameters over time in patients who have completed treatment for stage I-III cervical cancer receiving psychosocial telephone counseling vs usual care.
* Correlate psychosocial measures with immunologic stance.

OUTLINE: This is a randomized, controlled, parallel-group study. Patients are randomized to 1 of 2 intervention arms.

* Arm I: Patients undergo psychosocial telephone counseling comprising 5 weekly sessions and a 1-month follow-up session to learn strategies for reducing stress.
* Arm II: Patients undergo usual care for approximately 4 months. All patients complete questionnaires and Quality of life assessment at baseline and at 4 months. They also undergo saliva and blood sample collections at baseline and at 4 months for neuroimmune studies.

PROJECTED ACCRUAL: A total of 50 patients will be accrued for this study.

ELIGIBILITY:
INCLUSION CRITERIA

Disease Characteristics:

* Diagnosis of cervical cancer between the past 3-15 months

  * Stage I-III disease
* Completed therapy for cervical cancer ≥ 1 month ago

  * Not receiving ongoing treatment
* More than 4 weeks since prior immunotherapy
* More than 30 days since prior investigational drugs
* No prior biological response modifier
* No concurrent corticosteroids
* No concurrent immunosuppressive therapy

Patient Characteristics:

* Resident of Orange, San Diego, or Imperial County in California
* English or Spanish speaking
* No serious acute or chronic illness
* Has access to a telephone

EXCLUSION CRITERIA

Disease Characteristics:

* Stage IV cervical carcinoma
* Have undergone previous treatment with a biological response modifier (inferferons, interleukins) or prior immunotherapy within four weeks of study enrollment
* Used investigational drugs within 30 days of execution of the informed consent
* Required corticosteroids or were under immune suppression for any reason including an organ allograft or HIV infection
* Patients with metastatic disease or ongoing treatment
* Any acute or chronic illness, including autoimmune states, as judged clinically significant by the investigators

Patient Characteristics:

* Non-English or Spanish speakers

Ages: 18 Years to 120 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-08-01 (Actual); Primary Completion 2005-12-31 (Actual); Study Completion 2007-06-30 (Actual)

PRIMARY OUTCOMES:
Change in quality of life measured by FACT-Cx | Baseline and 4 months after enrollment
  FACT-Cx (Functional Assessment of Cancer Therapy-Cervical)
Change in neuroendocrine parameters | Baseline and 4 months after enrollment
  Saliva samples were tested for cortisol
Change in neuroendocrine parameters | Baseline and 4 months after enrollment
  Saliva samples were tested for dehydroepiandrosterone (DHEA) to calculate cortisol/DHEA ratios
Change in immune parameters | Baseline and 4 months after enrollment
  Blood samples were tested for T helper type 1and 2 (Th1/Th2) bias, as measured by IFN-γ/interleukin-5 ELISpot T
Change in immune parameters | Baseline and 4 months after enrollment
  Blood samples were tested for counterregulatory cytokine IL-10
Correlation of psychosocial measures and immunologic stance | Baseline and 4 months after enrollment
  Spearman's correlation coefficient between the change in FACT-Cx and the change in Th1/Th2 Immune system bias

CONTACTS AND LOCATIONS:
Overall Officials: Lari B. Wenzel, PhD, Principal Investigator — Chao Family Comprehensive Cancer Center
Locations (1):
- UCI, Health Policy and Research Center, Irvine, California, United States